CLINICAL TRIAL: NCT01340339
Title: Efficacy of Reverse Phototherapy With Super Light-emitting Diode(Super-led) in Term and Late Preterm Infants:Randomized and Controlled Clinical Trial
Brief Title: Reverse Phototherapy With Super Light-emitting Diode(Super-LED) for Hyperbilirubinemia in Term and Late Preterm Infants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Responsible Party: Danielle Cintra Bezerra Brandão, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FernandoFigueiraIMI
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: Jaundice; Hyperbilirubinemia; Phototherapy and Super-LED Fluorescent lamps
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Jaundice; Hyperbilirubinemia | interventions — Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BILITRON BED® (Experimental): Super-LED reverse phototherapy
  Interventions: Device: Phototherapy
- BILIBERÇO® (Active Comparator): Fluorescent Reverse Phototherapy
  Interventions: Device: Phototherapy

INTERVENTIONS:
Device: Phototherapy — Fluorescent reverse phototherapy (7 white lights 5cm below the base of acrylic cot), with spectral irradiance of 8-12microwatts/cm2/nm; daily; until bilirubin reaches level that indicates suspension of therapy
  Other Names: Fluorescent Light reverse phototherapy
  Arms: BILIBERÇO®
Device: Phototherapy — super LED reverse phototherapy (17 bulbs arranged in 42 x 31 cm in blue base acrylic cot), with spectral irradiance of 8-12microwatts/cm2/nm; daily; until bilirubin reaches level that indicates suspension of therapy
  Other Names: Super-LED reverse phototherapy
  Arms: BILITRON BED®

SUMMARY:
The aim of this study is to compare the efficacy of super-LED reverse phototherapy with the fluorescent reverse phototherapy in term and late preterm newborns.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial with hospitalized infants in the Professor Fernando Figueira Medicine Institute(IMIP), who require phototherapy as an indication of the medical team. Following the sample calculation, 144 patients will be randomized according to gestational age (350/7-376/7 or 380/7-416/7 weeks) to receive super-LED reverse phototherapy or fluorescent reverse phototherapy with spectral irradiance of 8-12 microwatts/cm2/nm.The bilirubin will be determined by micromethod with bilirubinometer, after blood collection in heparinized capillary until bilirubin reaches level that indicates suspension of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Newborns in the maternity Professor Fernando Figueira Medicine Institute(IMIP)
* Gestational age between 350/7 and 416/7 weeks
* Birth weight greater than 2200g
* Absence of congenital malformations
* indication of phototherapy after 48 hours of life
* Terms of consent signed by parent or guardian

Exclusion Criteria:

* Total Bilirubin level indicative of phototherapy intensive or exchange transfusion
* RH incompatibility hemolytic disease
* Mother's refusal to continue to participate in the study
* Unavailability of the two types of phototherapy equipment for randomization
* Mother or newborn who received phenobarbital

Ages: 35 Weeks to 41 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-10 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Bilirubinemia | 24 hours
  Bilirubin seric level decrease after 24 hours of phototherapy

SECONDARY OUTCOMES:
Phototherapy Time | 24 to 48 hours
  Number of hours needed to achieve a sufficiently low level of bilirubin that may allow suspension of phototherapy according to gestational age protocol.
Adverse Effects | 24 to 48 hours
  If any of the following are presented: weight loss, hypothermia or hyperthermia and/or skin lesions
Treatment Cost | 24 to 48 hours
  number of lamps exchanges needed to maintain necessary irradiance
Treatment Failure | 24 to 48 hours
  In cases in which increase in irradiance(>30microwatts/cm2/nm) is needed to lower bilirubin levels.
Rebound Hyperbilirubinemia | 24 hours
  Increased bilirubin seric levels, after suspension of phototherapy, with clinical necessity of phototherapy restart.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Brandão, Principal Investigator — Professor Fernando Figueira Medicine Institute
Locations (1):
- Danielle Cintra Bezerra Brandão, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Brandao DC, Draque CM, Sanudo A, de Gusmao Filho FA, de Almeida MF. LED versus daylight phototherapy at low irradiance in newborns >/=35 weeks of gestation: randomized controlled trial. J Matern Fetal Neonatal Med. 2015;28(14):1725-30. doi: 10.3109/14767058.2014.966678. Epub 2014 Nov 5. PMID 25234100